CLINICAL TRIAL: NCT05149599
Title: Efficacy and Safety of Saccharomyces Cerevisiae for Abdominal Pain and Discomfort in Irritable Bowel Syndrome (IBS) Patients
Brief Title: Saccharomyces Cerevisiae for Irritable Bowel Syndrome
Acronym: IBS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ziauddin University (Other)
Collaborators: Hilton Pharma (Industry)
Responsible Party: Principal Investigator, DR MEHREEN SIYAL, Resident Gastroenterology, Ziauddin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2731020MSGE
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated patients (Experimental)
  Interventions: Drug: Saccharomyces cerevisiae

INTERVENTIONS:
Drug: Saccharomyces cerevisiae — Saccharomyces cerevisiae, which is a pro-biotic, was given in capsule form, 500mg twice daily for 1 month

SUMMARY:
This study is designed to see the response of saccharomyces cerevisiae for symptomatic improvement of patients with IBS

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 75 years of age,
* Patients having confirmed IBS according to Rome IV criteria (newly and previously non-responder to treatment),
* Pain/ discomfort score strictly above 1 and strictly below 6 as determined on a pain/ discomfort scale using arbitrary grading from 0 to 7 in 7 days preceding the inclusion visit,
* Not hypersensitive to any of the ingredients of the drug.

Exclusion Criteria:

* Patients with an organic intestinal disease (Crohn's disease, ulcerative colitis, etc.),
* Pregnant females
* Treatments likely to influence IBS (anti-depressants, opioids, and narcotic analgesics)
* Patients with chronic alcoholism, vegetarian or vegan regimens
* Eating disorders such as anorexia or bulimia
* Documented food allergies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
To determine the response of saccharomyces cerevisiae for symptomatic improvement in patients with Irritablebowel syndrome through pain/ discomfort score | One month
  Responders were defined as the patients who had an improvement of 50% of the weekly average intestinal pain/discomfort score compared with the baseline average score for at least 2 out of the 4 weeks of study duration

SECONDARY OUTCOMES:
To determine the response of saccharomyces cerevisiae for symptomatic improvement in patients with IBS through IBS quality of life questionnaire | One month
  The IBS-QOL was evaluated using a validated 34-item IBS-QOL questionnaire, with each item scored on a 5-point Likert response scale (1 = not at all, 2 = slightly, 3 = moderately, 4 = quite a bit, and 5 = 'extremely' or 'a great deal'). The individual responses to the 34 items of the IBS-QOL questionnaire were summed and averaged for a total score and then transformed to a 0-100 scale for ease of interpretation, with higher scores indicating better IBS specific quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mehreen Siyal, MBBS, FCPS-1, Principal Investigator — DR ZIAUDDIN HOSPITAL, CLIFTON CAMPUS
Locations (1):
- Dr. Ziauddin University Hospital Clifton, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No